CLINICAL TRIAL: NCT07116707
Title: Effectiveness of Teacher-led Mental Health Literacy Programs on Knowledge, Stigma, and Help-seeking in Preteens: A Cluster Randomized Controlled Trial
Brief Title: Teacher-led MHL Education in Japanese Preteens
Acronym: SMHLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Nobuko Demura, Principal Investigator (PhD Student), Graduate School of Education, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SMHLP-JP-2019; 15H03083 (Other Grant/Funding Number: Japan Society for the Promotion of Science)
Record Dates: First submitted 2025-08-06; First posted 2025-08-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Literacy; Stigma of Mental Illness; Help-Seeking Behavior
Keywords: Mental Health Literacy; Stigma; Help-Seeking; Preteens; Elementary School Students; School-Based Intervention; Teacher-Led Program; Cluster Randomized Controlled Trial; Education Program; Japan
MeSH Terms: conditions — Help-Seeking Behavior; Social Stigma

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with school-level randomization.
Masking Description: Although classroom teachers may have been aware of group assignment, participants (students) were not informed of the study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teacher-Led Mental Health Literacy (MHL) Group (Experimental): Students in this group received a 45-minute mental health literacy (MHL) lesson led by their homeroom teacher. The session included three components: a slide-based introduction to mental health, a 10-minute animated video showing a student experiencing psychological stress, and a reflection activity using a worksheet. Teachers prepared for the lesson using self-guided materials, including a manual and instructional videos.
  Interventions: Behavioral: Short Mental Health Literacy Program (SMHLP)
- Waitlist Control Group (No Intervention): Students in this group received the standard school curriculum and did not receive the mental health literacy (MHL) lesson during the study period. The MHL lesson was provided to this group after the follow-up data collection for ethical reasons, but the post-lesson data were not included in the analysis.

INTERVENTIONS:
Behavioral: Short Mental Health Literacy Program (SMHLP) — A single 45-minute behavioral health education lesson delivered by homeroom teachers. The session included a slide-based introduction to mental health, a 10-minute animated video about a student experiencing psychological stress, and a worksheet-based reflection activity. Teachers prepared using self-guided materials.
  Arms: Teacher-Led Mental Health Literacy (MHL) Group

SUMMARY:
The goal of this clinical trial is to learn whether a short, teacher-delivered mental health literacy (MHL) program can help improve mental health knowledge, reduce stigma, and encourage help-seeking among preteens in Japan. Participants are students in grade 5 (age 10-11) and grade 6 (age 11-12) attending public elementary schools.

The main questions this study aims to answer are:

* Does the program increase students' knowledge about mental health and illnesses?
* Does it reduce stigma toward people with mental illnesses?
* Does it increase willingness to seek help and support peers?

Researchers will compare students who receive the program with those who follow the usual school curriculum.

Participants will:

* Answer short self-report questionnaires before, right after, and three months after the program
* Learn through a 45-minute classroom session that includes slides, a short animated film, and review activities
* Be part of regular school classes led by their homeroom teacher

The goal is to understand whether a concise and scalable MHL education can support early mental health awareness and prevention in younger youth.

The results may help schools provide effective mental health education at an early age.

DETAILED DESCRIPTION:
This study used a cluster randomized controlled trial design, with randomization at the school level. Eight public elementary schools in Kanazawa City were assigned to either intervention or control groups using simple randomization by external staff not involved in implementation.

The intervention, the Short Mental Health Literacy Program (SMHLP), consisted of a 45-minute classroom lesson delivered by homeroom teachers. The lesson included three parts: a slide-based introduction to mental health, a 10-minute original animation about a student experiencing psychological stress, and a worksheet-based reflection activity. Teachers used self-guided materials including videos and manuals to prepare.

Primary outcome measures included an 8-item true/false knowledge scale (range: 0-8), a 5-item social distance scale (range: 5-20), and binary-response questions on help-seeking intention and willingness to support peers. The internal consistency of the knowledge scale was acceptable (Cronbach's α = 0.65), and that of the stigma scale was good (Cronbach's α = 0.88).

Data were collected at three time points: before the intervention (T1), immediately after (T2), and three months later (T3). **Statistical analyses were conducted using linear mixed models (LMM) for continuous outcomes and logistic regression mixed models (LRMM) for binary outcomes. Three-level hierarchical structures were modeled for LMM, with time nested within students and students nested within schools. School-level clustering was adopted. For LRMMs, two-level models were used without random effects for schools due to convergence issues. Intention-to-treat analyses were conducted.** Subgroup analyses were performed by grade level.

Parental opt-out consent procedures were used, and verbal assent was obtained from students. The study was approved by the University of Tokyo Human Research Ethics Committee (Approval No. 15-118).

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in 5th or 6th grade at one of the eight participating public elementary schools in Kanazawa, Japan.
* Aged 10-12 years old.
* Passive consent obtained from guardians; verbal assent obtained from children.
* Able to complete self-report questionnaires.

Exclusion Criteria:

* Students whose parents/guardians opted out of the study.

Note: Students who were absent on the day of the pre-test (T1) were excluded from the analysis population but not from the initial study cohort.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1401 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mental Health Knowledge Score | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  An 8-item true/false questionnaire developed based on the SMHLP content. Scores range from 0 to 8, with higher scores indicating greater knowledge about mental health and illnesses. Cronbach's alpha was 0.65.

SECONDARY OUTCOMES:
Social Distance Scale Score (Stigma) | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  A 5-item scale adapted from the Social Distance Scale using a vignette format. Each item rated on a 4-point scale (1=definitely willing to 4=definitely unwilling), total score range 4-20. Higher scores indicate greater stigma. Cronbach's alpha was 0.88.
Help-Seeking Intention | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  A vignette-based item asking whether students themselves would seek help if they were experiencing similar mental health difficulties. Responses were on a 4-point scale: "Definitely yes", "Probably yes", "Probably not", and "Definitely not". Students were considered to have the intention to seek help if they responded "Definitely yes".
Recognition of the necessity to seek help | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  A single vignette-based item asking whether students thought the character in the scenario should seek help from others. Responses were on a 4-point scale: "Definitely yes", "Probably yes", "Probably not", and "Definitely not". Students were considered to recognize the necessity to seek help when they responded "Definitely yes".
Intention to Help Peers | Baseline (T1), immediately post-intervention (T2), and 3-month follow-up (T3)
  Students were asked to rate their likelihood of performing various desirable supportive behaviors for a peer in distress. Each item was rated on a 4-point scale. Students were considered to have the intention to help if they selected "Definitely yes" for at least one of the behaviors. An example of a behavior is: "I would ask about or listen to their story to understand their situation in detail."

CONTACTS AND LOCATIONS:
Locations (1):
- Kanazawa Municipal Elementary Schools (8 schools), Kanazawa, Ishikawa-ken, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be made available upon request. The final decision on data sharing will be made in consultation with the principal investigator.
Supporting Information: SAP
Time Frame: Data may become available beginning 6 months following publication and up to 36 months after publication, pending approval by the principal investigator.
Access Criteria: Access to the data may be granted to qualified researchers affiliated with academic institutions for secondary analyses. Requests will be reviewed by the research team in consultation with the principal investigator to ensure ethical and legal compliance.